CLINICAL TRIAL: NCT01776749
Title: Subcutaneous Stimulation as Add on Therapy to Spinal Cord Stimulation (SCS) to Treat Low Back Pain in Failed Back Surgery Syndrome (FBSS) (SubQ Study)
Brief Title: Subcutaneous Stimulation as Add on Therapy to SCS toTreat Low Back Pain in FBSS
Acronym: SubQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SubQ (Other)
Collaborators: Radboud University Medical Center (Other); Albert Schweitzer Hospital (Other); Maastricht University Medical Center (Other); Rijnstate Hospital (Other); Rijnland Hospital (Other); Medtronic (Industry); Sint Maartenskliniek (Other); Diakonessenhuis locatie Zeist (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL324.091.10
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Low Back Pain; Failed Back Surgery Syndrome; Neuropathic Pain
Keywords: low back pain; failed back surgery syndrome; spinal cord stimulation; subcutaneous stimulation; peripheral nerve field stimulation
MeSH Terms: conditions — Low Back Pain; Failed Back Surgery Syndrome; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- no SubQ (No Intervention): No subcutaneous leads due to adequate low back stimulation by only SCS. Patient not randomised
- SubQ ON (Active Comparator): Subcutaneous stimulation on
  Interventions: Device: SubQ
- SubQ OFF (Sham Comparator): subcutaneous leads implanted, but no stimulation
  Interventions: Device: SubQ

INTERVENTIONS:
Device: SubQ — Spinal Cord Stimulation (SCS) and subcutaneous (SubQ) stimulation SCS trial stimulation: Implantation of the Octad lead in the epidural space. The lead implantation in the epidural space is performed under local anesthesia using a standard percutaneous technique. A key element to the technical success of an SCS procedure is the accurate placement of the lead, which results in paresthesia covering the patients' painful areas. This depends on the patients' feedback during intra-operative testing. Therefore, it is important that the patient is awake and fully cooperative during the trial stimulation.
  Other Names: The octad lead (3877)SubQ leads (3888); (Prime Advanced 37702 or Restore Advanced 37713); all Medtronic
  Arms: SubQ OFF; SubQ ON

SUMMARY:
Aim of the study Failed back surgery syndrome (FBSS) is a clinical entity consisting of chronic leg and /or back pain due to radicular nerve damage. The effectiveness of Spinal Cord Stimulation (SCS) in the pain management of patients with FBSS is proven. Patients mostly have dominant leg pain, however a significant percentage of FBSS patients has a more pronounced back pain and are commonly excluded from SCS as it is often inadequate in relieving both the back and leg pain components. Recently some reports showed the benefit of subcutaneous stimulation (SubQ) for low back pain in patients with FBSS. This has been confirmed by a feasibility study performed by our group. The aim of the randomized controlled study is to evaluate the effect of SubQ on low back pain in FBSS patients for whom SCS gives an inadequate back pain relief.

Hypothesis We hypothesize that SubQ in addition to SCS in FBSS patients with leg and low back pain is more effective in treating low back pain (i.e. >50% pain reduction) than SCS alone.

DETAILED DESCRIPTION:
Aim of the study FBSS is a clinical entity consisting of chronic leg and /or back pain due to radicular nerve damage. The effectiveness of SCS in the pain management of patients with FBSS is proven. Patients mostly have dominant leg pain, however a significant percentage of FBSS patients has a more pronounced back pain and are commonly excluded from SCS as it is often inadequate in relieving both the back and leg pain components. Recently some reports showed the benefit of subcutaneous stimulation (SubQ) for low back pain in patients with FBSS. This has been confirmed by a feasibility study performed by our group. The aim of the randomized controlled study is to evaluate the effect of SubQ on low back pain in FBSS patients for whom SCS gives an inadequate back pain relief.

Hypothesis We hypothesize that SubQ in addition to SCS in FBSS patients with leg and low back pain is more effective in treating low back pain (i.e. >50% pain reduction) than SCS alone.

Study design and duration of the study The study is a randomized controlled trial. Patients with FBSS with additional chronic back pain and an intensity of 5 or more for leg and back pain separately on the visual analogue scale are eligible for the study. About ninety patients will receive a SCS system targeting to relief leg and back pain. The study group consists of patients having a pain reduction of ≥50% in the leg after SCS trial stimulation. If, after trial stimulation, there is less than 50% back pain relief compared with initial values, patients will receive one or two Quad leads subcutaneously at the time of implantation of the pulse generator.

This group, a total of 56 patients,will be randomized in a 1:1 ratio in which group 1 (n=28) receives SCS plus non-activated SubQ(SubQ OFF) and group 2 (n=28) receives SCS plus activated SubQ (SubQ ON) (phase 1), for a period of 3 months.

After the controlled phase of the study, all 56 patients will receive maximal effective SCS and SubQ for the rest of the study duration (phase 2).

Total duration of the study for a patient is12 months. Estimated duration of the study is 18 months.

Comparisons will be made after 3 months between no SubQ OFF and SubQ ON. After 6 and 12 months (phase 2) patients will be compared with their baseline values to explore long term effects of SCS and SubQ.

Type and number of patients The study will include FBSS patients with leg and low back pain, failing to relief back pain with SCS. For the controlled part of the study 56 patients are needed based on a power calculation in which a difference between the two treatments is postulated of about 40%. To assure this about 90 patients will be included in the study.

Inclusion criteria Male/female > 18 and < 75 years Chronic neuropathic pain secondary to FBSS Pain radiating in lumbar segments L4 and/or L5 and/or S1 for at least 6 months Pain intensity assessed by VAS ≥ 5 scored separately for leg and back Willing to provide informed consent Exclusion criteria Presence of any other clinically significant or disabling chronic pain condition Expected inability of patients to properly operate the neurostimulation system History of coagulation disorders, lupus erythematosus, diabetes mellitus, rheumatoid arthritis or morbus Bechterew Active malignancy Current use of medicines affecting coagulation which cannot be temporarily stopped Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator Life expectancy of less than 1 year Existing or planned pregnancy Study therapy test therapy: Adequate subcutaneous stimulation with perceived paresthesias in the painful area in the back reference therapy: SCS plus non-activated SubQ (SubQ OFF) Parameters for evaluation of effectiveness primary outcome: The proportion of patients with SCS plus activated SubQ and SCS without activated SubQ having 50% or more pain relief(responder rate) in back after 3 months of stimulation, assessed with the VAS.

secondary outcomes:

Effect of SCS plus activated SubQ and SCS without activated SubQ after 3, 6 and 12 months on:

Mean reduction in pain intensity for leg and back pain separately, assessed by the VAS Responder rate of SCS on leg pain assessed by the VAS Responder rate of SubQ on back pain assessed by the VAS(after 6 and 12 months) Quality of life assessed by Short Form 36 (SF-36) Quality of life as assessed by EuroQuol (EQ-5D) Function assessed by the Oswestry disability index Patient satisfaction assessed by the Global Impression of Change (GPIC) Pain assessed by the McGill questionnaire Concomitant drug treatment for relief of pain Concomitant need for physical therapy or other non-drug treatment. Employment status Frequency and nature of adverse events

And in addition after 12 months of stimulation, on:

Cost-utility Preferred stimulation settings

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Chronic pain secondary to FBSS. Pain radiating in lumbar segments L4 and/or L5 and/or S1 for at least 6 months following at least one anatomically successful surgery.
* Pain intensity in leg(s) and low back of 5 or higher for leg and back measured separately on a weighted visual analogue scale (VAS).
* Previous treatment has been unsuccessful (insufficient pain relief and/or unacceptable side-effects).
* Willing to provide informed consent.

Exclusion Criteria:

* Exclusion criteria
* Presence of any other clinically significant or disabling chronic pain condition
* Expected inability of the patient to properly operate the neurostimulation system
* History of coagulation disorders, lupus erythematosus, diabetes mellitus, rheumatoid arthritis or morbus Bechterew
* Current use of medication affecting coagulation which cannot be temporarily stopped
* Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact the perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by the investigator
* The patient has ever had SCS
* Addiction: drugs, alcohol (>5 U / day) and/or medication
* Insufficient cooperation from the patient (little motivation, understanding or communication)
* Immune deficiency (HIV-positive, corticosteroids with a dose equivalent to

  * prednisolone 10 mg, immunosuppressives, etc.)
* Life expectancy < 1 year
* Pacemaker
* Local infection or other skin disorders at site of incision
* Existing or planned pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11-09 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2015-07-11 (Actual)

PRIMARY OUTCOMES:
responder rate | 3 months
  The proportion of patients with SCS plus activated SubQ and SCS without activated SubQ having 50% or more pain relief(responder rate) in back after 3 months of stimulation, assessed with the VAS

CONTACTS AND LOCATIONS:
Overall Officials: Kris CP Vissers, MD,PhD,FIPP, Study Chair — Radboud University Medical Center; Eric-Jan JA van Gorp, MD, Principal Investigator — Albert Schweitzer Hospital
Locations (1):
- Albert Schweitzer hospital, Dordrecht, South Holland, Netherlands

REFERENCES:
- [Derived] van Heteren EPZ, van Roosendaal BWP, van Gorp EJAA, Bronkhorst EM, Kallewaard JW, Wegener JT, Burger K, Teernstra OPM, Buschman HPJ, Hamm-Faber TE, Vissers KCP. Spinal Cord Stimulation With Additional Peripheral Nerve/Field Stimulation Versus Spinal Cord Stimulation Alone on Back Pain and Quality of Life in Patients With Persistent Spinal Pain Syndrome. Neuromodulation. 2023 Apr;26(3):658-665. doi: 10.1016/j.neurom.2021.11.010. Epub 2022 Jan 26. PMID 35088732